CLINICAL TRIAL: NCT04302753
Title: Autistic Women's Experiences of Self Compassion and Receiving Their Diagnosis in Adulthood
Status: Completed | Type: Observational
Sponsor: University of Sheffield (Other)
Responsible Party: Sponsor
Other Study IDs: 164845
Record Dates: First submitted 2020-02-13; First posted 2020-03-10 (Actual); Last update posted 2021-05-06 (Actual); Status verified 2020-03

CONDITIONS: Autism
Keywords: Autism; Self compassion
MeSH Terms: conditions — Autistic Disorder

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Research highlights strong links between self-compassion and mental health, but there is very limited research specifically exploring autistic individual's experiences of self-compassion. The process of receiving a diagnosis on the autism spectrum can be complex and autistic women tend to experience several barriers to diagnosis. This study adds to the growing area of research exploring autistic women's experiences of receiving a diagnosis in adulthood. This study employs Interpretative phenomenological analysis to explore if receiving a diagnosis of Autism influences women's perceptions of self-compassion. The findings may inform client-centred practices in health care settings and potentially present positive aspects of autism diagnosis.

ELIGIBILITY:
Inclusion Criteria:

* Able to consent to participate
* Cisgender female (female at birth and raised as female).
* Speak English fluently
* Received an Autism Spectrum Disorder diagnosis, aged 18 years old or above

Exclusion Criteria:

* Lack capacity to consent to participate in the study
* Unable to speak English fluently
* Have not received an Autism diagnosis
* Have received Autism diagnosis prior to their 18th birthday
* Have an intellectual disability
* Born male

Ages: 18 Years to 99 Years | Sex: Female
Age Groups: Adult, Older Adult
Gender Based: Yes — To be cisgender female (female at birth and raised as female).
Study Population: Women who have received their diagnosis on the autism spectrum over the age of 18 years old.
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2019-08-12 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2021-03-29 (Actual)

PRIMARY OUTCOMES:
Experience of receiving ASD diagnosis in adulthood based on semi structured interviews | day one
  Participants' experience of receiving ASD diagnosis in adulthood based on semi structured interviews, completed in one interview.

SECONDARY OUTCOMES:
Experience of self-compassion before and after receiving ASD diagnosis based on semi structured interviews | day one
  Participants' experiences of self-compassion before and after receiving ASD diagnosis based on semi structured interviews, completed in one interview.

CONTACTS AND LOCATIONS:
Locations (1):
- DClin Univeristy of Sheffield, Sheffield, Yorkshire and Humber, United Kingdom

IPD SHARING:
Plan to Share IPD: No
All electronic data including transcripts and audio recordings will be stored in the university data repository, until publication and dissemination of the study is completed. The paper copies of anonymized interview transcripts will be stored in a locked cabinet in the research administration office at the university of Sheffield, for a maximum of six years and then destroyed confidentially.